CLINICAL TRIAL: NCT00004978
Title: A Randomized, Open-Label, Phase III, International Study of Subcutaneous Recombinant IL-2 in Patients With HIV-1 Infection and CD4+ Cell Counts 300/mm^3 or Greater: Evaluation of Subcutaneous Proleukin in a Randomized International Trial
Brief Title: An International Study to Evaluate Recombinant Interleukin-2 in HIV Positive Patients Taking Anti-retroviral Therapy
Acronym: ESPRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPRIT 001; 5U01AI046957 (NIH); 00 I-0071; 3U01AI046957-05S2 (NIH); 3U01AI046957-05S3 (NIH); 10118 (Registry Identifier: DAIDS ES Registry Number); NCT00004737 (obsolete NCT alias)
Record Dates: First submitted 2000-03-10; First posted 2001-08-31 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Injections, Subcutaneous; HIV-1; Interleukin-2; Drug Therapy, Combination; CD4 Lymphocyte Count; Disease Progression; Follow-Up Studies; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Disease Progression | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rIL-2 (Experimental): Recombinant interleukin-2 (rIL-2) therapy used with combination anti-HIV medication of choice.
  Interventions: Drug: Recombinant interleukin-2 (rIL-2)
- No rIL-2 (No Intervention): Control arm uses anti-HIV medication of choice without rIL-2.

INTERVENTIONS:
Drug: Recombinant interleukin-2 (rIL-2) — Recombinant interleukin-2 at a dose of 7.5 MIU given twice daily subcutaneously for 5 consecutive days every 8 weeks for at least 3 cycles.
  Other Names: Proleukin; IL-2; Aldesleukin
  Arms: rIL-2

SUMMARY:
The purpose of this study is to see if it is effective to give HIV positive patients recombinant interleukin-2 (rIL-2) in addition to anti-HIV therapy. Patients will be followed over a minimum of 4 years to study the long-term effects of rIL-2 on their HIV disease progression.

Anti-HIV therapy has been very successful in treating HIV positive patients and in keeping viral load (level of HIV in the blood) low. However, anti-HIV drugs cannot completely rid the body of the virus, and the immune system is never completely restored in HIV positive patients. Doctors hope that giving patients recombinant interleukin-2 (rIL-2) in addition to their anti-HIV therapy will help improve their immune systems and keep them healthier over a longer period of time. rIL-2 is a hormone naturally produced by the body during an immune response to a microbial infection.

DETAILED DESCRIPTION:
Much progress has been made in implementing potent antiretroviral therapy that is able to maximally suppress viral replication. However, these drug combinations do not result in viral eradication and, for many patients, virologic and immunologic control cannot be maintained. Even among patients with apparent virologic control, a "ceiling effect" seems to exist with failure of CD4 cell counts to rise on average more than 100 to 150 cells/mm^3, at least during the first 2 years of therapy. The incomplete recovery of immune function after initiation of therapy remains an obstacle in the management of HIV. Preservation of immune function by direct expansion of CD4 lymphocytes with rIL-2 could represent a significant additional treatment strategy. It also has been speculated recently that rIL-2 in combination with potent antiretroviral therapy may be a useful approach for purging HIV from the latently infected CD4 cells. It is hoped that intervention with rIL-2 therapy in combination with antiretroviral therapy at an early stage of HIV infection can prevent CD4 T-cell depletion and result in fewer AIDS-defining illnesses than with antiretroviral therapy alone.

Patients are randomized to receive subcutaneous (SC) rIL-2 therapy or no rIL-2 therapy. All patients must be taking a regimen of combination antiretroviral treatment, with the choice of therapy at the discretion of the treating clinician. Antiretroviral medications are not provided by this study. Recombinant IL-2 is given SC for 5 consecutive days every 8 weeks for at least 3 cycles unless toxicities or other contraindications develop. After the first three cycles, additional cycles are given at the discretion of each patient's physician, with a general goal of maintaining the patient's CD4 cell count at twice the baseline level or at 1,000 cells/mm^3 or above for as long as possible. Patients in the no rIL-2 group receive no injections. Patients in both treatment groups are seen every 4 months for follow-up data collection to monitor viral load and CD4 cell counts. All patients are followed for a minimum of 4 years. During the trial, patients in the no SC rIL-2 group are not given rIL-2 at any point. However, at the end of the study, if rIL-2 is found to be effective in reducing the rate of disease progression [AS PER AMENDMENT 12/15/00: (new and recurrent events)], including death, all patients are offered rIL-2.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Have a CD4 cell count of 300 cells/mm3 or more within 45 days of study entry
* Are on combination anti-HIV therapy or are beginning anti-HIV therapy at the time of study entry
* Are at least 18 years old

Exclusion Criteria:

* Have received IL-2 before
* Have cancer requiring chemotherapy
* Have evidence of active clinical disease within the past year for any AIDS-defining illness or certain other conditions such as herpes zoster or Chagas disease. (This study has been changed. Previously, patients were ineligible if they had a history of any AIDS-defining illness or certain other conditions.)
* Have used certain medications, such as corticosteroids or drugs affecting the immune system, in the 45 days before study entry
* Have a nervous system disorder requiring antiseizure medication
* Have an autoimmune or inflammatory disease such as inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), psoriasis, optic neuritis, or any autoimmune/inflammatory diseases with potentially life-threatening complications
* Are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4150 (Actual)
Dates: Start 2000-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Abrams, MD, Study Chair — University of California, San Francisco; Marcelo Losso, MD, Study Chair — Hospital Jose Maria Ramos Mejia, Buenos Aires, Argentina
Locations (248):
- United States (78):
  - VA Greater Los Angeles Healthcare System, Infectious Diseases Section CRS, Los Angeles, California
  - Dr. M. Estes Med. Practice CRS, Mill Valley, California
  - Dr. Robert Scott Med. Practice CRS, Oakland, California
  - East Bay AIDS Ctr. CRS, Oakland, California
  - Dr. Shawn Hassler Med. Practice CRS, San Francisco, California
  - Positive Health Program Clinic (San Francisco Gen. Hosp.) CRS, San Francisco, California
  - Positive Health Practice West/ Dr. Steve Deeks CRS, San Francisco, California
  - Dr. William Owen Med. Practice CRS, San Francisco, California
  - Dr. Martin Mass Med. Practice CRS, San Francisco, California
  - San Francisco VAMC, Infectious Diseases Clinic CRS, San Francisco, California
  - UCSF PHP, Gen. Internal Medicine Practice CRS, San Francisco, California
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - Dr. Virginia Cafaro Med. Practice CRS, San Francisco, California
  - Denver Infectious Diseases Consultants CRS, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Whitman-Walker Clinic CRS, Washington D.C., District of Columbia
  - George Washington Univ. Med. Ctr. Infectious Diseases - Clinical Trials Unit CRS, Washington D.C., District of Columbia
  - Walter Reed Army Med. Ctr., Infectious Disease Clinic CRS, Washington D.C., District of Columbia
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Dr. Timothy A. Price Med. Practice CRS, Washington D.C., District of Columbia
  - Miami VAMC CRS, Miami, Florida
  - Univ. of Miami, Infectious Diseases Clinical Research Unit CRS, Miami, Florida
  - ARCA, Central Clinc CRS, Atlanta, Georgia
  - Emory Univ. Crawford Long Hosp. CRS, Atlanta, Georgia
  - Atlanta VAMC CRS, Decatur, Georgia
  - Klein & Slotten Medical Associates CRS, Chicago, Illinois
  - Jesse Brown VAMC CRS, Chicago, Illinois
  - Univ. of Illinois Family Ctr. for Infectious Disease CRS, Chicago, Illinois
  - Lakeshore Infectious Disease Associates CRS, Chicago, Illinois
  - North Side Family Medicine CRS, Chicago, Illinois
  - Northwestern Memorial Physicians Group CRS, Chicago, Illinois
  - Med. Ctr. of Louisiana at New Orleans, HIV Outpatient Clinics CRS, New Orleans, Louisiana
  - Tulane University Health Sciences Center, Louisiana Community AIDS Research Program(LaCARP) CRS, New Orleans, Louisiana
  - New Orleans VAMC CRS, New Orleans, Louisiana
  - NIH Clinical Ctr., NIAID HIV Clinic CRS, Bethesda, Maryland
  - National Naval Med. Ctr., Infectious Diseases Special Immunology Clinic CRS, Bethesda, Maryland
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Wayne State Univ. CRS, Detroit, Michigan
  - St. John Hosp. & Med. Ctr., Infectious Diseases Dept. CRS, Grosse Pointe Woods, Michigan
  - William Beaumont Hosp., Infectious Disease Research CRS, Royal Oak, Michigan
  - Abbott Northwestern Hosp., Clinic 42 CRS, Minneapolis, Minnesota
  - Mayo Clinic INSIGHT CRS, Rochester, Minnesota
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - ID Care Inc. - Hillsborough CRS, Hillsborough, New Jersey
  - Jersey Shore Univ. Med. Ctr. CRS, Neptune City, New Jersey
  - New Jersey Community Research Initiative, Jeffrey Bomser Clinic CRS, Newark, New Jersey
  - Cathedral Healthcare System, St. Michael's Med. Ctr. CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey CRS, Paterson, New Jersey
  - Raritan Bay Med. Ctr., Perth Amboy Division CRS, Perth Amboy, New Jersey
  - ID Care - Randolph CRS, Randolph Township, New Jersey
  - Infectious Disease Specialists of N.J., North Jersey Community Research Initiative CRS, Union, New Jersey
  - The Early Intervention Program at Kennedy Hosp. CRS, Voorhees Township, New Jersey
  - St. Vincent Hosp. & Med. Ctr. CRS, New York, New York
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Jacobi Med. Ctr., Ambulatory Care Pavillion CRS, The Bronx, New York
  - Bronx VAMC CRS, The Bronx, New York
  - Oregon Health & Sciences Univ. Internal Medicine (L-475) CRS, Portland, Oregon
  - Multnomah County Health Dept., HIV Health Services Ctr. CRS, Portland, Oregon
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Providence Portland Med. Ctr., Ambulatory Care and Education Ctr. CRS, Portland, Oregon
  - Kaiser Immune Deficiency Clinic of Portland CRS, Portland, Oregon
  - Legacy Clinic Emanuel CRS, Portland, Oregon
  - Salem Hosp. CRS, Salem, Oregon
  - Kaiser Permanente Lancaster Clinic CRS, Salem, Oregon
  - Temple Univ. School of Medicine CRS, Philadelphia, Pennsylvania
  - Michael E. DeBakey VAMC CRS, Houston, Texas
  - Northwest Clinic CRS, Houston, Texas
  - Thomas Street Clinic CRS, Houston, Texas
  - Univ. Clinical Research Ctr., Memorial Hermann Hosp. CRS, Houston, Texas
  - Legacy Community Health Services, Inc., Montrose Clinic, Inc., Houston, Texas
  - South Texas Veterans Health Care System, Immunosuppression Clinic CRS, San Antonio, Texas
  - Hanover Med. Park (Mechanicsville, VA) CRS, Mechanicsville, Virginia
  - Naval Med. Ctr. Portsmouth CRS, Portsmouth, Virginia
  - CrossOver Health Ctr. CRS, Richmond, Virginia
  - South Richmond Health Care Ctr. CRS, Richmond, Virginia
  - Hunter Holmes McGuire VAMC CRS, Richmond, Virginia
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
- Argentina (13):
  - Hosp. de Clinicas Jose de San Martin, Div. Infectologia CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hosp. Italiano de Buenos Aires, Infectious Diseases Section CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hosp. Gen. de Agudos JM Ramos Mejia, Servicio de Inmunocomprometidos CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hospital de Infecciosas F.J. Muniz CRS, Ciudad de Buenos Aires, Buenos Aires
  - Funcei Crs, Ciudad de Buenos Aires, Buenos Aires
  - Hosp. Gen. de Agudos Juan A. Fernandez CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hosp. Gen. de Agudos 'Teodoro Alvarez' CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hospital Nacional Professor Alejandro Posadas CRS, El Palomar, Buenos Aires
  - Hospital Interzonal de Agudos Oscar Alende, Sala de Infectologia CRS, Mar del Plata, Buenos Aires
  - Caici Crs, Rosario, Santa Fe Province
  - Hosp. Rawson CRS, Córdoba
  - Hosp. Interzonal de Agudos San Juan de Dios CRS, La Plata
  - Hosp. Central, Immunology Dept. CRS, Mendoza
- Australia (23):
  - Interchange General Practice CRS, Canberra, Australian Capital Territory
  - Canberra Hosp., Canberra Sexual Health Clinic CRS, Woden, Australian Capital Territory
  - Burwood Road Gen. Practice CRS, Burwood, New South Wales
  - St. Vincent's Hospital CRS, Darlinghurst, New South Wales
  - Taylor Square Private Clinic CRS, Darlinghurst, New South Wales
  - Holdsworth House Gen. Practice CRS, Darlinghurst, New South Wales
  - John Hunter Hosp., Immunology & Infectious Diseases Unit CRS, Newcastle, New South Wales
  - 407 Doctors CRS, Surry Hills, New South Wales
  - Albion Street Ctr. CRS, Surry Hills, New South Wales
  - Queensland Health - AIDS Med. Unit CRS, Brisbane, Queensland
  - Cairns Base Hosp., Sexual Health Services CRS, Cairns, Queensland
  - Gladstone Road Medical Ctr. CRS, Highgate Hill, Queensland
  - Nambour Gen. Hosp. CRS, Nambour, Queensland
  - Royal Adelaide Hosp. CRS, Adelaide, South Australia
  - The Care & Prevention Programme CRS, Adelaide, South Australia
  - Carlton Clinic CRS, Carlton, Victoria
  - The Alfred Hosp., Clinical Research - Infectious Diseases Unit CRS, Melbourne, Victoria
  - Prahran Market Clinic CRS, Melbourne, Victoria
  - Northcote Clinic CRS, Northcote, Victoria
  - Royal Melbourne Hosp., Victorian Infectious Diseases Service CRS, Parkville, Victoria
  - The Ctr. Clinic INSIGHT CRS, St Kilda, Victoria
  - Royal Perth Hospital CRS, Perth, Western Australia
  - Gold Coast Sexual Health Clinic CRS, Miami, Queensland
- Austria (2):
  - Univ. of Vienna Med. School, Div. of Allergy, Immunology & Infectious Diseases - Sued B CRS, Vienna
  - SMZ Baumgartner Hoehe, Immunambulanz Pavillion Wienerwald Parterre CRS, Vienna
- Ctr. Hospitalier Universitaire, St Pierre, Div. of Infectious Diseases (PL5) CRS, Brussels, Belgium
- Brazil (3):
  - Centro de Referencia e Treinamento em DST/AIDS - Sao Paulo CRS, Vila Mariana, São Paulo
  - Instituto de Infectologia Emilio Ribas CRS, São Paulo
  - Universidade Federal de Sao Paulo,IDIPA-Instituto Paulista de Doencas Infecciosas e Parasitarias CRS, São Paulo
- Canada (15):
  - Univ. of Alberta Hosp., Clinical Research Office CRS, Edmonton, Alberta
  - Cool Aid Community Health Ctr. CRS, Victoria, British Columbia
  - Q.E. II Health Sciences Ctr., Captial District Authority, Victoria Gen. Hosp. CRS, Halifax, Nova Scotia
  - The HAVEN Program, Sudbury Regional Hosp., Laurentian Site CRS, Greater Sudbury, Ontario
  - McMaster Univ. Med. Ctr. Hamiton Health Sciences, SIS Clinic CRS, Hamilton, Ontario
  - St. Joseph's Health Ctr. of London, HIV Care Programme CRS, London, Ontario
  - Ottawa Hosp., Gen. Campus CRS, Ottawa, Ontario
  - Toronto Gen. Hosp. Infectious Diseases CRS, Toronto, Ontario
  - Windsor Regional Hosp., HIV Care Program CRS, Windsor, Ontario
  - CHUS - Hopital Fleurimont, Centre de Recherche Clinique CRS, Fleurimont, Quebec
  - Hopital Maisonneuve-Rosemont, Dept. de Microbiologie CRS, Montreal, Quebec
  - CHUM - Campus Notre-Dame CRS, Montreal, Quebec
  - Royal Victoria Hosp., Montreal Chest Institute CRS, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec - CHUL, Centre de Recherche en Indectiologie CRS, Sainte-Foy, Quebec
  - Royal Univ. Hosp. CRS, Saskatoon, Saskatchewan
- Denmark (5):
  - Aalborg Hosp., Dept. of Infectious Diseases CRS, Aalborg
  - Skejby Sygehus, Department of Infectious Diseases Q (ambulatoriet) CRS, Aarhus
  - Rigshospitalet, Department of Infectious Diseases, M5112 CRS, Copenhagen
  - Hvidovre Univ. Hosp., Dept. of Infectious Diseases CRS, Hvidovre
  - Odense Univ. Hosp., Med. Dept. C CRS, Odense
- France (22):
  - Centre Hospitalier de la Region Annecienne, Service des Maladie Infectieuses CRS, Cedex, Pringy
  - CHRU d'Angers, Service de Maladies Infectieuses CRS, Angers
  - Hopital Saint-Jacques, Service des Maladies Infectieuses et Tropicales CRS, Besançon
  - Hopital Avicenne, Service de Medecine B CRS, Bobigny
  - Hopital Antoine Beclere Service d'Immunologie Clinique CRS, Clamart
  - Hopital Louis Mourier, Service de Medecine Interne CRS, Colombes
  - Hopital Henri Mondor, Immunopathologie Clinique CRS, Créteil
  - Hopital Raymond Poincare - Vidal 2, Service des Maladies Infectieuses et Tropicales CRS, Garches
  - Hopital de Bicetre, Service de Medecine Interne CRS, Le Kremlin-Bicêtre
  - Hopital Sainte Marguerite, CISIH Hopital de Jour CRS, Marseille
  - Hopital de la Conception, Service des Maladies Infectieuses CRS, Marseille
  - Hopital Gui de Chauliac, Service des Maladies Infectieuses et Tropicales CRS, Montpellier
  - Hopital de l'Archet 1, Service de Medecine Interne 2 Hematologie Clinique CRS, Nice
  - Hopital Saint-Antoine, Service de Maladies Infectieuses CRS, Paris
  - Hopital de La Salpetriere, Service de Medecine Interne CRS, Paris
  - Hopital Cochin, Service de Medecine Interne 2 CRS, Paris
  - Hopital Necker, Service des Maladies Infectieuses CRS, Paris
  - Hopital Europeen Georges Pompidou, Service d'Immunologie Clinique CRS, Paris
  - Hopital Tenon, Service de Maladies Infectieuses et Tropicales CRS, Paris
  - C.H.U. Bichat - Claude Bernard Service des Maladies Infectieuses et Tropicales CRS, Paris
  - CHRU de Strasbourg (France) CRS, Strasbourg
  - Hopital Foch, Service de Medecine Interne CRS, Suresenes
- Germany (10):
  - Univ. Hosp. Charite, Dept of Infectious Diseases CRS, Berlin
  - Ruhr-Univ., Interdiszipl. Immunolog. Ambulanz CRS, Bochum
  - Medizinische Universitaetsklinik - Bonn, Immunologische Ambulanz CRS, Bonn
  - Klinik I fur Innere Medizin der Universitat zu Koln, Studienburo fur Infektiologie u. HIV CRS, Cologne
  - Ctr. for HIV & Hepatogastroenterology, HIV Specialised Practice (Private Practice) CRS, Düsseldorf
  - Johann Wolfgang Goethe Univ. Hosp., Infektionsambulanz CRS, Frankfurt
  - IPM Study Ctr. (Hamburg) CRS, Hamburg
  - Univ. Hosp. Heidelberg, Dept. of Dermatology CRS, Heidelberg
  - Klinikum Innenstadt, Infektionsambulanz und Tagesklinik CRS, München
  - Univ. of Wuerzburg, Medizinische Poliklinik, Schwerpunkt Hepatologie/Infektiologie CRS, Würzburg
- St. James' Hosp., Guide Clinic CRS, Dublin, Ireland
- Israel (3):
  - Rambam Med. Ctr., Immunology, Allergy & AIDS Institute, B. Rappaport Faculty of Medicine, Technion, Haifa
  - Kaplan Med. Ctr., Ben Ari Institute of Clinical Immunology CRS, Rehovot
  - Tel Aviv Sourasky Med. Ctr., Clinical Immunology Unit and AIDS Ctr. CRS, Tel Aviv
- Italy (8):
  - Civili di Brescia, 1st Division of Infectious Diseases CRS, Brescia
  - Civili di Brescia, Dept of Infectious & Tropical Disease, Hosp.Spedali Civili of Brescia CRS, Brescia
  - Ospedale S. Maria Annunziata, U.O. Malattie Infettive CRS, Florence
  - Ospedale San Raffaele, Centro San Luigi - Divisione Malattie Infettive CRS, Milan
  - Univ. of Milan, Ospedale Luigi Sacco, Institute of Infectious and Tropical Diseases CRS, Milan
  - Universita degli Studi di Modena e Reggio Emilia, Clinica delle Malattie Infettive e Tropicali CRS, Modena
  - San Matteo Hospital - University of Pavia, Division of Infectious and Tropical Diseases CRS, Pavia
  - Universita La Sapienza, Clinica Universita La Sapienza CRS, Roma
- Japan (3):
  - Osaka National Hosp. AIDS Ctr., Clinical Research Institute CRS, Osaka
  - International Med. Ctr. of Japan CRS, Tokyo
  - Univ. of Tokyo, Research Hosp. of the Institute of Medical Science CRS, Tokyo
- Univ. Hosp. Ctr. of the Med. School of Casablanca, Infectious Diseases Unit CRS, Casablanca, Morocco
- Netherlands (6):
  - OLVG -- locatie Prinsengracht, Dept. of Internal Medicine II CRS, Amsterdam
  - Academisch Medisch Centrum CRS, Amsterdam
  - Stichting Medisch Centrum Jan van Goyen, Dept. of Internal Medicine CRS, Amsterdam
  - Groningen Univ. Hosp., Department of Internal Medicine CRS, Groningen
  - Kennemer Gasthuis, Lokatie EG CRS, Haarlem
  - St. Elisabeth Ziekenhuis CRS, Tilburg
- Ulleval Hosp., Dept. of Infectious Diseases CRS, Oslo, Norway
- Poland (4):
  - Szpital Specjalistyczny, Osrodek Diagnostyki i Terapii AIDS CRS, Chorzów
  - Pomeranian Academy of Medicine (PAM), Dept. of Infectious Diseases and Hepatology CRS, Szczecin
  - Wojewodzki Szpital Zakazny CRS, Warsaw
  - Wroclaw Univ., School of Med., Dept. of Infectious Diseases, Liver Diseases and AIDS CRS, Wroclaw
- Portugal (3):
  - Hospital de Cascais, HDDI, Departamento Medicina Interna CRS, Cascais
  - Hosp. de Egas Moniz, Servicio de Infecciologia e Medicina Tropical CRS, Lisbon
  - Hosp. de Santa Maria, Servico de Doencas Infecciosas CRS, Lisbon
- Tan Tock Seng Hosp., Infectious Diseases Research Ctr. CRS, Singapore, Singapore
- Spain (17):
  - Hosp. Donostia CRS, Donostia / San Sebastian, Guipuzcoa
  - Hosp. Juan Canalejo, Dept. of Internal Medicine CRS, A Coruña
  - Hosp. Santa Creu i Sant Pau, Servicio de Medicina Interna CRS, Barcelona
  - Hosp. Clinico de Barcelona CRS, Barcelona
  - Hosp. del Mar, Internal Medicine-Infectious Diseases CRS, Barcelona
  - Hosp. Universitari Germans Trias i Pujol, HIV Unit and Retrovirology Lab. CRS, Barcelona
  - Hosp. Universitario Gregorio Maranion, Microbiology & Infectious Diseases Unit CRS, Madrid
  - Centro de Investigacion Carlos III, Infectious Diseases Dept. CRS, Madrid
  - Hosp. Severo Ochoa, Internal Medicine and Infectious Diseases CRS, Madrid
  - Hosp. 12 de Octubre, Pabellon de Medicina Communitaria CRS, Madrid
  - Hosp. Clinico San Carlos CRS, Madrid
  - Hosp. la Princesa, Internal Medicine and Infectious Diseases Service CRS, Madrid
  - Hosp. Ramon y Cajal (Madrid) CRS, Madrid
  - Hosp. Universitario La Paz CRS, Madrid
  - Hosp. Universitario Principe de Asturias CRS, Madrid
  - Hosp. Universitario Morales Meseguer CRS, Murcia
  - Hosp. Virgen del Rocio, Infectious Diseases Service CRS, Seville
- Sweden (2):
  - Karolinska Univ. Hosp. Huddinge, Dept. of Infectious Diseases CRS, Stockholm
  - Venhalsan, Soder Hosp., Dept. of Infectious Diseases, Karolinska Univ. Hosp. CRS, Stockholm
- Regional Hosp. of Lugano (Sede Civico), Ospedale Civico di Lugano, Infectious Diseases Unit CRS, Lugano, Canton Ticino, Switzerland
- Thailand (5):
  - Siriraj Hosp., Mahidol Univ. INSIGHT CRS, Bangkok, Ratchathewi
  - Chulalongkorn Univ. Hosp., HIV-NAT Research Collaboration CRS, Bangkok, Ratchathewi
  - Chiang Rai Regional Hosp. INSIGHT CRS, Chiangrai
  - Chonburi Regional Hosp., Dept. of Internal Medicine CRS, Chon Buri
  - Khon Kaen Univ., Srinagarind Hosp., Div. of Infectious Diseases & Tropical Medicine, Dept. of Medici, Khon Kaen
- United Kingdom (20):
  - Brighton & Sussex Univ. Hosp. NHS Trust, HIV Research Office CRS, Elm Grove, Brighton
  - Royal Victoria Hosp. Dept. of Genitourinary Medicine CRS, Belfast, Northern Ireland
  - Churchill Hosp. John Warin Ward CRS, Headington, Oxford
  - Western Gen. Hosp., Regional Infectious Diseases Unit CRS, Edinburgh, Scotland
  - Gartnaval Gen. Hosp., Brownlee Ctr. CRS, Glasgow, Scotland
  - Heartlands Hosp. Dept. of Infection & Tropical Disease Outpatients CRS, Birmingham
  - Royal Devon & Exeter NHS Foundation Trust, Heavitree Hosp., Dept. of GU Medicine CRS, Exeter
  - Leicester Royal Infirmary, Dept. of Infection & Tropical Medicine CRS, Leicester
  - Royal London Hosp., Ambrose King Ctr. CRS, London
  - St. Thomas' Hosp., Dept. of GU Medicine CRS, London
  - St. George's Hosp. Clinical Infection UnitCRS, London
  - Chelsea & Westminster Hosp., St. Stephens Ctr. CRS, London
  - King's College Hosp., Caldecot Ctr. Dept. of Sexual Health CRS, London
  - Royal Free Hosp., Dept. of Infection & Immunity, Ian Charleson Day Ctr. CRS, London
  - St. Bartholomew's Hosp., Infection & Immunity Clinical Group CRS, London
  - St. Mary's Hosp. of London, Imperial College School of Medicine CRS, London
  - Univ. College London Med. School, Ctr. for Sexual Health & HIV Research CRS, London
  - Newcastle Gen. Hosp., Dept of Infection & Tropical Medicine CRS, Newcastle upon Tyne
  - Edith Cavell Hosp. Dept. of Sexual Health, Clinic E CRS, Peterborough
  - Royal Hallamshire Hosp., Dept. of GU Medicine Communicable Diseases Unit CRS, Sheffield

REFERENCES:
- [Background] Chun TW, Engel D, Mizell SB, Hallahan CW, Fischette M, Park S, Davey RT Jr, Dybul M, Kovacs JA, Metcalf JA, Mican JM, Berrey MM, Corey L, Lane HC, Fauci AS. Effect of interleukin-2 on the pool of latently infected, resting CD4+ T cells in HIV-1-infected patients receiving highly active anti-retroviral therapy. Nat Med. 1999 Jun;5(6):651-5. doi: 10.1038/9498. PMID 10371503
- [Background] Connors M, Kovacs JA, Krevat S, Gea-Banacloche JC, Sneller MC, Flanigan M, Metcalf JA, Walker RE, Falloon J, Baseler M, Feuerstein I, Masur H, Lane HC. HIV infection induces changes in CD4+ T-cell phenotype and depletions within the CD4+ T-cell repertoire that are not immediately restored by antiviral or immune-based therapies. Nat Med. 1997 May;3(5):533-40. doi: 10.1038/nm0597-533. PMID 9142122
- [Background] Emery S, Abrams DI, Cooper DA, Darbyshire JH, Lane HC, Lundgren JD, Neaton JD; ESPRIT Study Group. The evaluation of subcutaneous proleukin (interleukin-2) in a randomized international trial: rationale, design, and methods of ESPRIT. Control Clin Trials. 2002 Apr;23(2):198-220. doi: 10.1016/s0197-2456(01)00179-9. PMID 11943448
- [Result] Arduino RC, Nannini EC, Rodriguez-Barradas M, Schrader S, Losso M, Ruxrungtham K, Allende MC, Emery S, Fosdick L, Neaton J, Tavel JA, Davey RT, Lane HC; Evaluation of Subcutaneous Proleukin in a Randomized International Trial (ESPRIT) Vanguard Group; ESPRIT Executive Committee. CD4 cell response to 3 doses of subcutaneous interleukin 2: meta-analysis of 3 Vanguard studies. Clin Infect Dis. 2004 Jul 1;39(1):115-22. doi: 10.1086/421775. Epub 2004 Jun 14. PMID 15206062
- [Result] INSIGHT-ESPRIT Study Group; SILCAAT Scientific Committee; Abrams D, Levy Y, Losso MH, Babiker A, Collins G, Cooper DA, Darbyshire J, Emery S, Fox L, Gordin F, Lane HC, Lundgren JD, Mitsuyasu R, Neaton JD, Phillips A, Routy JP, Tambussi G, Wentworth D. Interleukin-2 therapy in patients with HIV infection. N Engl J Med. 2009 Oct 15;361(16):1548-59. doi: 10.1056/NEJMoa0903175. PMID 19828532
- [Derived] Larson GS, Carey C, Grarup J, Hudson F, Sachi K, Vjecha MJ, Gordin F; INSIGHT Group. Lessons learned: Infrastructure development and financial management for large, publicly funded, international trials. Clin Trials. 2016 Apr;13(2):127-36. doi: 10.1177/1740774515625974. Epub 2016 Feb 8. PMID 26908541
- [Derived] Nordell AD, McKenna M, Borges AH, Duprez D, Neuhaus J, Neaton JD; INSIGHT SMART, ESPRIT Study Groups; SILCAAT Scientific Committee. Severity of cardiovascular disease outcomes among patients with HIV is related to markers of inflammation and coagulation. J Am Heart Assoc. 2014 May 28;3(3):e000844. doi: 10.1161/JAHA.114.000844. PMID 24870935
- [Derived] Mocroft A, Neuhaus J, Peters L, Ryom L, Bickel M, Grint D, Koirala J, Szymczak A, Lundgren J, Ross MJ, Wyatt CM; INSIGHT SMART Study Group; ESPRIT Study Group. Hepatitis B and C co-infection are independent predictors of progressive kidney disease in HIV-positive, antiretroviral-treated adults. PLoS One. 2012;7(7):e40245. doi: 10.1371/journal.pone.0040245. Epub 2012 Jul 20. PMID 22911697
- [Derived] Pett SL, Carey C, Lin E, Wentworth D, Lazovski J, Miro JM, Gordin F, Angus B, Rodriguez-Barradas M, Rubio R, Tambussi G, Cooper DA, Emery S; INSIGHT-ESPRIT Study Group. Predictors of bacterial pneumonia in Evaluation of Subcutaneous Interleukin-2 in a Randomized International Trial (ESPRIT). HIV Med. 2011 Apr;12(4):219-27. doi: 10.1111/j.1468-1293.2010.00875.x. Epub 2010 Aug 31. PMID 20812949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled to ESPRIT between 2000 and 2003. As per the ESPRIT protocol, patients from previous Vanguard studies (in Thailand, Argentina, and the U.S., enrolled 1997-1999) were followed and included in the analysis cohort of this study if at least 90% of patients from that site consented to ESPRIT.
Groups:
- rIL-2: Subcutaneous recombinant interleukin-2 (rIL-2) therapy
- No rIL-2: Control group - no study-assigned medication
Period: Overall Study
Arm/Group | rIL-2 | No rIL-2
Started | 2090 (includes patients participating in Vanguard studies from the sites which participated in ESPRIT) | 2060 (includes patients participating in Vanguard studies from the sites which participated in ESPRIT)
Completed | 1846 | 1790
Not Completed | 244 | 270
Not completed — Death | 107 | 116
Not completed — Lost to Follow-up | 101 | 108
Not completed — Withdrawal by Subject | 17 | 26
Not completed — site closure - not in analysis cohort | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rIL-2 | No rIL-2 | Total
Number analyzed (Participants) | 2090 | 2060 | 4150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2071 | 2032 | 4103
  >=65 years | 19 | 28 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (8.8) | 40.9 (9.1) | 40.8 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 388 | 381 | 769
  Male | 1702 | 1679 | 3381
Region of Enrollment [Number; unit: participants]
  Argentina | 276 | 278 | 554
  Australia | 107 | 98 | 205
  Austria | 16 | 18 | 34
  Belgium | 39 | 41 | 80
  Brazil | 48 | 50 | 98
  Canada | 74 | 67 | 141
  Denmark | 39 | 33 | 72
  France | 86 | 96 | 182
  Germany | 136 | 130 | 266
  Ireland | 3 | 1 | 4
  Israel | 31 | 33 | 64
  Italy | 50 | 54 | 104
  Japan | 14 | 11 | 25
  Morocco | 12 | 14 | 26
  Netherlands | 29 | 25 | 54
  Norway | 3 | 5 | 8
  Poland | 48 | 52 | 100
  Portugal | 51 | 56 | 107
  Singapore | 10 | 10 | 20
  Spain | 151 | 157 | 308
  Sweden | 4 | 3 | 7
  Switzerland | 5 | 5 | 10
  Thailand | 182 | 183 | 365
  United Kingdom | 165 | 163 | 328
  United States | 511 | 477 | 988
CD4+ cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 465 [374 to 592] | 451 [370 to 578] | 458 [373 to 586]

OUTCOME MEASURES:

1. Primary Outcome: New or Recurrent HIV Disease Progression Event Including Death
Description: Participants who die or experience at least one: any CDC Category C 1993 AIDS-defining events or one of the following: invasive aspergillosis, bartonellosis, Chagas disease, Herpes zoster, visceral Leishmaniasis, Hodgkin's lymphoma, non-Hodgkin's lymphoma (all cell types), microsporidiosis, nocardiosis, disseminated Penicillium marneffii, extrapulmonary Pneumocystis carinii, and Rhodococcus equi disease
Time Frame: from randomization through study end - median of 7.6 years follow-up
Population: ITT
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
participants | 159 | 165
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .55, Regression, Cox — P-value is 2-sided using an alpha of .05; Hazard ratio is from unadjusted proportional hazards regression model; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.16] — HR is for rIL-2 vs control

2. Secondary Outcome: New or Recurrent Serious HIV Disease Progression Event Including Death
Description: Patients with at least one: progressive multifocal leukoencephalopathy, lymphoma, visceral Kaposi's sarcoma, AIDS dementia complex, toxoplasmosis, histoplasmosis, cryptococcosis, Mycobacterium avium complex, wasting syndrome, and cytomegalovirus disease.
Time Frame: from randomization through study end - median of 7.6 years follow-up
Population: ITT
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
participants | 126 | 130
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .62, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.74 to 1.20]

3. Secondary Outcome: Number of Participants Who Died From Any Cause
Time Frame: from randomization through study end - median of 7.6 years follow-up
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
participants | 107 | 116
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .42, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.69 to 1.17]

4. Secondary Outcome: Participants With a New Disease Progression Event or Death
Description: Includes first new episode of: CDC Category C 1993 AIDS-defining events plus invasive aspergillosis, bartonellosis, Chagas disease, Herpes zoster, visceral Leishmaniasis, Hodgkin's lymphoma, non-Hodgkin's lymphoma (all cell types), microsporidiosis, nocardiosis, disseminated Penicillium marneffii, extrapulmonary Pneumocystis carinii, and Rhodococcus equi disease
Time Frame: from randomization through 15 November 2008 - median of 7.6 years follow-up
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
participants | 154 | 164
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .41, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.14]

5. Secondary Outcome: Absolute CD4 Cell Counts Averaged Throughout Followup
Description: Average of all available CD4+ cell counts measured at follow-up visits
Time Frame: from randomization through study end - median of 7.6 years follow-up
Population: CD4+ cell counts averaged over all participants with at least one CD4+ measurement recorded during follow-up.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2053 | 2024
cells/mm^3 | 715.4 (273.1) | 556.3 (193.0)
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; Mean Difference (Final Values) = 159, 95% CI 2-sided [145 to 174] — treatment difference (rIL2 - no rIL2) estimated from a longitudinal model that considers CD4+ measured at followup visits

6. Secondary Outcome: Plasma HIV RNA Levels
Description: log10 HIV-RNA averaged throughout follow-up
Time Frame: From randomization through study end - median of 7.6 years follow-up
Population: HIV-RNA measurement averaged over followup visits for all participants with at least one follow-up measurement.
Measure: Mean (Standard Deviation); unit: log10 HIV-RNA
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2065 | 2036
log10 HIV-RNA | 2.20 (0.65) | 2.17 (0.61)

7. Secondary Outcome: Number of Participants With Changes in Anti-retroviral Treatment (ART)
Description: Number of participants who changed ART at least once during the study period.
Time Frame: From randomization through study end - median of 7.6 years follow-up
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
participants | 1760 | 1751
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .07, Regression, Cox; Hazard ratio (rIL-2 vs. no rIL-2) for first change in antiretroviral treatment; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.88 to 1.00]

8. Secondary Outcome: Grade 4 Signs and Symptoms
Description: Participants with at least one grade 4 sign or symptom (except those limited to a laboratory measurement), other than AIDS-defining conditions. Events were graded according to a standardized toxicity table. Events not specifically contained in the toxicity table were considered Grade 4 if they resulted in extreme limitation in activity or required significant medical intervention/therapy, hospitalization or hospice care. Grade 4 events by type are given under the adverse events section.
Time Frame: From randomization through study end - median of 7.6 years follow-up
Measure: Number; unit: Participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
Participants | 466 | 383
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .003, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [1.07 to 1.41] — HR (IL-2 vs control) for first grade 4 event, ITT analysis

9. Secondary Outcome: Pattern of Use of Prophylaxis for Opportunistic Infections
Description: Number of participants using pneumocystis pneumonia (PCP) prophylaxis at the last attended followup visit.
Time Frame: last followup visit - median of 7.6 years follow-up
Population: Intention to treat (ITT) - Medication use recorded on the last followup visit attended among all participants attending at least one followup visit.
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2028 | 2005
participants | 54 | 53
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .97, Chi-squared

10. Secondary Outcome: Hepatic, Metabolic, and Cardiac Conditions
Description: Number of participants experiencing a "serious non-AIDS" event defined as first serious cardiovascular, renal, or hepatic event, or non-AIDS malignancy.
Time Frame: From randomization through study end - median of 7.6 years follow-up
Measure: Number; unit: participants
Arm/Group | rIL-2 | No rIL-2
Number analyzed (Participants) | 2071 | 2040
participants | 134 | 136
Statistical Analysis 1: Comparison: rIL-2 vs No rIL-2; Test type: Superiority or Other; p = .74, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.76 to 1.22]

ADVERSE EVENTS:
Time Frame: Grade 4 events were reportable from randomization through study end (15 November 2008), irrespective of whether patient was taking a study treatment.
Description: Adverse events are grade 4 events (excluding AIDS-defining events and events limited to abnormal laboratory values), reportable in both treatment arms. All grade 4 events are included under "serious adverse events", categorized according to MedDRA HLGT. Common adverse events of any grade are reported under "other adverse events" by MedDRA PT.
Arm/Group | rIL-2 | No rIL-2
Serious Adverse Events (participants affected / at risk) | 466/2071 | 383/2040
Other Adverse Events (participants affected / at risk) | 133/2071 | 92/2040
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rIL-2 (N=2071) | No rIL-2 (N=2040)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 7 | 9
Platelet disorders (Blood and lymphatic system disorders) | 1 | 3
Spleen, lymphatic, and reticuloendothelial system disorders (Blood and lymphatic system disorders) | 3 | 1
White blood cell disorders (Blood and lymphatic system disorders) | 0 | 5
cardiac arrhythmias (Cardiac disorders) | 6 | 4
cardiac valve disorders (Cardiac disorders) | 3 | 0
Coronary artery disorders (Cardiac disorders) | 41 | 46
Heart failures (Cardiac disorders) | 6 | 0
Myocardial disorders (Cardiac disorders) | 0 | 2
Pericardial disorders (Cardiac disorders) | 2 | 1
Inner ear and VIIIth cranial nerve disorders (Ear and labyrinth disorders) | 2 | 0
Middle ear disorders (excl congenital) (Ear and labyrinth disorders) | 1 | 0
Adrenal gland disorders (Endocrine disorders) | 1 | 0
Thyroid gland disorders (Endocrine disorders) | 5 | 2
Ocular infections, irritations and inflammations (Eye disorders) | 2 | 0
Ocular neuromuscular disorders (Eye disorders) | 0 | 1
Ocular structural change, deposit and degeneration NEC (Eye disorders) | 1 | 2
Vision disorders (Eye disorders) | 1 | 0
Abdominal hernias and other abdominal wall conditions (Gastrointestinal disorders) | 3 | 6
Anal and rectal conditions NEC (Gastrointestinal disorders) | 1 | 5
Benign neoplasms gastrointestinal (Gastrointestinal disorders) | 1 | 0
Diverticular disorders (Gastrointestinal disorders) | 1 | 1
Exocrine pancreas conditions (Gastrointestinal disorders) | 8 | 11
Gastrointestinal conditions NEC (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhages NEC (Gastrointestinal disorders) | 8 | 9
Gastrointestinal inflammatory conditions (Gastrointestinal disorders) | 1 | 3
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 11 | 9
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 15 | 13
Gastrointestinal stenosis and obstruction (Gastrointestinal disorders) | 2 | 2
Gastrointestinal ulceration and perforation (Gastrointestinal disorders) | 5 | 1
Gastrointestinal vascular conditions (Gastrointestinal disorders) | 2 | 2
Peritoneal and retroperitoneal conditions (Gastrointestinal disorders) | 0 | 3
Administration site reactions (General disorders) | 0 | 1
Body temperature conditions (General disorders) | 15 | 4
General system disorders NEC (General disorders) | 17 | 6
Therapeutic and nontherapeutic effects (excl toxicity) (General disorders) | 1 | 0
Tissue disorders NEC (General disorders) | 2 | 0
Bile duct disorders (Hepatobiliary disorders) | 3 | 1
Gallbladder disorders (Hepatobiliary disorders) | 10 | 10
Hepatic and hepatobiliary disorders (Hepatobiliary disorders) | 13 | 8
Allergic conditions (Immune system disorders) | 3 | 2
Immune disorders NEC (Immune system disorders) | 1 | 1
Bacterial infectious disorders (Infections and infestations) | 20 | 17
Fungal infectious disorders (Infections and infestations) | 3 | 0
Infections - pathogen unspecified (Infections and infestations) | 47 | 42
Mycobacterial infectious disorders (Infections and infestations) | 1 | 1
Protozoal infectious disorders (Infections and infestations) | 0 | 1
Viral infectious disorders (Infections and infestations) | 19 | 18
Bone and joint injuries (Injury, poisoning and procedural complications) | 15 | 8
Chemical injury and poisoning (Injury, poisoning and procedural complications) | 4 | 4
Injuries NEC (Injury, poisoning and procedural complications) | 9 | 13
Medication errors (Injury, poisoning and procedural complications) | 5 | 1
Procedural and device related injuries and complications NEC (Injury, poisoning and procedural complications) | 1 | 1
Enzyme investigations NEC (Investigations) | 1 | 0
Gastrointestinal investigations (Investigations) | 1 | 0
Haematology investigations (incl blood groups) (Investigations) | 1 | 3
Hepatobiliary investigations (Investigations) | 6 | 1
Lipid analyses (Investigations) | 1 | 0
Metabolic, nutritional and blood gas investigations (Investigations) | 1 | 0
Physical examination topics (Investigations) | 2 | 0
Renal and urinary tract investigations and urinalyses (Investigations) | 1 | 0
Acid-base disorders (Metabolism and nutrition disorders) | 3 | 3
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 2 | 4
Glucose metabolism disorders (incl diabetes mellitus) (Metabolism and nutrition disorders) | 6 | 5
Lipid metabolism disorders (Metabolism and nutrition disorders) | 2 | 0
Bone disorders (excl congenital and fractures) (Musculoskeletal and connective tissue disorders) | 3 | 5
Connective tissue disorders (excl congenital) (Musculoskeletal and connective tissue disorders) | 1 | 0
Fractures (Musculoskeletal and connective tissue disorders) | 3 | 0
Joint disorders (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle disorders (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal and connective tissue deformities (incl intervertebral disc disorders) (Musculoskeletal and connective tissue disorders) | 2 | 5
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 2 | 6
Synovial and bursal disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast neoplasms malignant and unspecified (incl nipple) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Endocrine neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Endocrine neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Gastrointestinal neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 8
Haematopoietic neoplasms (excl leukaemias and lymphomas) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatic and biliary neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatobiliary neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Leukaemias (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Miscellaneous and site unspecified neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Miscellaneous and site unspecified neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9
Renal and urinary tract neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Reproductive neoplasms female benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Reproductive neoplasms female malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Reproductive neoplasms male malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Respiratory and mediastinal neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 8
Skin neoplasms malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 4
Soft tissue neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Central nervous system infections and inflammations (Nervous system disorders) | 1 | 0
Central nervous system vascular disorders (Nervous system disorders) | 16 | 11
Cranial nerve disorders (excl neoplasms) (Nervous system disorders) | 2 | 0
Demyelinating disorders (Nervous system disorders) | 1 | 0
Encephalopathies (Nervous system disorders) | 1 | 2
Headaches (Nervous system disorders) | 5 | 6
Increased intracranial pressure and hydrocephalus (Nervous system disorders) | 1 | 0
Movement disorders (incl parkinsonism) (Nervous system disorders) | 3 | 0
Neurological disorders NEC (Nervous system disorders) | 9 | 12
Neuromuscular disorders (Nervous system disorders) | 2 | 0
Peripheral neuropathies (Nervous system disorders) | 2 | 4
Seizures (incl subtypes) (Nervous system disorders) | 8 | 4
Spinal cord and nerve root disorders (Nervous system disorders) | 1 | 0
Structural brain disorders (Nervous system disorders) | 1 | 1
Abortions and stillbirth (Pregnancy, puerperium and perinatal conditions) | 3 | 1
Foetal complications (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Maternal complications of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Postpartum and puerperal disorders (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety disorders and symptoms (Psychiatric disorders) | 4 | 1
Deliria (incl confusion) (Psychiatric disorders) | 0 | 1
Depressed mood disorders and disturbances (Psychiatric disorders) | 13 | 9
Disturbances in thinking and perception (Psychiatric disorders) | 1 | 0
Eating disorders and disturbances (Psychiatric disorders) | 0 | 1
Impulse control disorders NEC (Psychiatric disorders) | 0 | 1
Manic and bipolar mood disorders and disturbances (Psychiatric disorders) | 2 | 0
Mood disorders and disturbances NEC (Psychiatric disorders) | 1 | 1
Personality disorders and disturbances in behaviour (Psychiatric disorders) | 0 | 1
Psychiatric disorders NEC (Psychiatric disorders) | 3 | 5
Schizophrenia and other psychotic disorders (Psychiatric disorders) | 4 | 3
Suicidal and self-injurious behaviours NEC (Psychiatric disorders) | 18 | 10
Bladder and bladder neck disorders (excl calculi) (Renal and urinary disorders) | 1 | 0
Nephropathies (Renal and urinary disorders) | 1 | 1
Renal disorders (excl nephropathies) (Renal and urinary disorders) | 9 | 10
Urethral disorders (excl calculi) (Renal and urinary disorders) | 1 | 0
Urinary tract signs and symptoms (Renal and urinary disorders) | 6 | 4
Urolithiases (Renal and urinary disorders) | 3 | 5
Breast disorders (Reproductive system and breast disorders) | 0 | 1
Cervix disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 2 | 3
Menstrual cycle and uterine bleeding disorders (Reproductive system and breast disorders) | 1 | 1
Ovarian and fallopian tube disorders (Reproductive system and breast disorders) | 1 | 0
Prostatic disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 1 | 0
Testicular and epididymal disorders (Reproductive system and breast disorders) | 1 | 1
Uterine, pelvic and broad ligament disorders (Reproductive system and breast disorders) | 3 | 1
Bronchial disorders (excl neoplasms) (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Lower respiratory tract disorders (excl obstruction and infection) (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pleural disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary vascular disorders (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Angioedema and urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 6 | 3
Skin and subcutaneous tissue disorders NEC (Skin and subcutaneous tissue disorders) | 1 | 0
Skin appendage conditions (Skin and subcutaneous tissue disorders) | 0 | 1
Skin vascular abnormalities (Social circumstances) | 0 | 1
Legal issues (Social circumstances) | 0 | 1
Hepatobiliary therapeutic procedures (Surgical and medical procedures) | 0 | 1
Obstetric and gynaecological therapeutic procedures (Surgical and medical procedures) | 0 | 2
Aneurysms and artery dissections (Vascular disorders) | 1 | 1
Arteriosclerosis, stenosis, vascular insufficiency and necrosis (Vascular disorders) | 6 | 2
Decreased and nonspecific blood pressure disorders and shock (Vascular disorders) | 5 | 0
Embolism and thrombosis (Vascular disorders) | 9 | 3
Vascular disorders NEC (Vascular disorders) | 2 | 0
Vascular haemorrhagic disorders (Vascular disorders) | 1 | 1
Vascular hypertensive disorders (Vascular disorders) | 6 | 3
Venous varices (Vascular disorders) | 0 | 1
Muscuoloskeletal and connective tissue disorders congenital (Congenital, familial and genetic disorders) | 1 | 0
Diabetic complications (Metabolism and nutrition disorders) | 1 | 0
Soft tissue sarcomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rIL-2 (N=2071) | No rIL-2 (N=2040)
Acute myocardial infarction (Cardiac disorders) | 16 | 15
Anaemia (Blood and lymphatic system disorders) | 9 | 10
Appendicitis (Infections and infestations) | 10 | 8
Cerebrovascular accident (Nervous system disorders) | 12 | 4
Coronary artery disease (Cardiac disorders) | 12 | 9
Deep vein thrombosis (Vascular disorders) | 10 | 2
Depression (Psychiatric disorders) | 14 | 7
Diarrhoea (Gastrointestinal disorders) | 16 | 10
Myocardial infarction (Cardiac disorders) | 14 | 18
Pyrexia (General disorders) | 18 | 9
Suicide attempt (Psychiatric disorders) | 11 | 10
Vomiting (Gastrointestinal disorders) | 13 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No